CLINICAL TRIAL: NCT00418405
Title: Hanyang University Medical Center Arthritis Network
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hanyang University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: HUMAN
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2007-01

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis, Rheumatoid; Cohort Studies
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Rheumatoid arthritis is a relatively common autoimmune disease that affects about 1% of the population. Its impact on health-related quality of life of the affected patients and the national medical cost are enormous. However, a systemic prospective cohort study of rheumatoid arthritis has not yet been established in Korea, so data on characteristics and prognosis of Korean rheumatoid arthritis and their response to therapy and adverse events are limited. Therefore establishment of large prospective cohort of Korean rheumatoid arthritis is imperative.

With inauguration of a steadfast prospective cohort of Korean rheumatoid arthritis patients in The Hospital for Rheumatic Diseases at Hanyang University, where patients gather from all over Korea forming the largest and most diverse patient pool in Korea, we will be able to define the characteristics and prognosis of Korean rheumatoid arthritis patients and gather information on treatment response and adverse events. This will eventually lead to improvement of health-related quality of life in Korean rheumatoid arthritis patients and provide opportunity for reliable comparison study with research institutes from other countries. The data gathered through the cohort will provide valuable foundational information for the genetic studies, pharmacological economic analyses, and standard treatment guidelines of Korean rheumatoid arthritis patients.

DETAILED DESCRIPTION:
This study is a longitudinal prospective cohort of Korean rheumatoid arthritis patients comprising of all Korean adult rheumatoid arthritis patients satisfying the 1987 revised American College of Rheumatology (ACR) criteria and voluntarily agreeing to participate in the study with following objectives;

Primary Objectives:

1. Gather information on treatment response and adverse events of various pharmacological therapies for treatment of Korean rheumatoid arthritis patients
2. Identify the incidence and mortality rates of concurrent diseases including the cardiovascular & gastrointestinal diseases and assess the contributing factors involved

Secondary Objectives:

Enrich understanding of disease characteristics, treatment response and adverse events in Korean rheumatoid arthritis to promote health and increase the health-related quality of life in Korean rheumatoid arthritis patients

ELIGIBILITY:
Inclusion Criteria:

* Korean adult rheumatoid arthritis patients satisfying the 1987 revised American College of Rheumatology (ACR) criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500
Dates: Start 2007-01; Study Completion 2012-01

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Cheol Bae, MD, PhD, MPH, Principal Investigator — Hanyang University
Locations (1):
- The Hospital for Rheumatic Diseases, Hanyang University, Seoul, South Korea